CLINICAL TRIAL: NCT05375838
Title: Phase 1/2, Randomized, Stratified, Observer-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1073 (SARS-CoV-2 and Influenza Vaccine) Compared to Co-administered mRNA-1010 (Influenza) and mRNA-1273 (SARS-CoV-2) Vaccines and to mRNA- 1010 Vaccine and mRNA-1273 Vaccine Alone in Healthy Adults 18-75 Years of Age
Brief Title: A Safety, Reactogenicity, and Immunogenicity Study of mRNA-1073 (COVID-19/Influenza) Vaccine in Adults 18 to 75 Years Old
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: mRNA-1073-P101
Record Dates: First submitted 2022-05-13; First posted 2022-05-17 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: SARS-CoV-2; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1073 COVID-19 and influenza combined vaccine; mRNA-1010 influenza vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- mRNA-1273 Plus Placebo (Experimental): Participants will receive 2 intramuscular (IM) injections, one in each arm, of mRNA-1273 plus placebo at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1273; Biological: Placebo
- mRNA-1010 Plus Placebo (Experimental): Participants will receive 2 IM injections, one in each arm, of mRNA-1010 plus placebo at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1010; Biological: Placebo
- mRNA-1010 Plus mRNA-1273 (Experimental): Participants will receive 2 IM injections, one in each arm, of mRNA-1010 plus mRNA-1273 at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1010
- Dose A: mRNA-1073 Plus Placebo (Experimental): Participants will receive 2 IM injections, one in each arm, of mRNA-1073 plus placebo at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1073; Biological: Placebo
- Dose B: mRNA-1073 Plus Placebo (Experimental): Participants will receive 2 IM injections, one in each arm, of mRNA-1073 plus placebo at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1073; Biological: Placebo
- Dose C: mRNA-1073 Plus Placebo (Experimental): Participants will receive 2 IM injections, one in each arm, of mRNA-1073 plus placebo at the specified dose level on Day 1.
  Interventions: Biological: mRNA-1073; Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1073 — Sterile liquid for injection
  Arms: Dose A: mRNA-1073 Plus Placebo; Dose B: mRNA-1073 Plus Placebo; Dose C: mRNA-1073 Plus Placebo
Biological: mRNA-1010 — Sterile liquid for injection
  Arms: mRNA-1010 Plus Placebo; mRNA-1010 Plus mRNA-1273
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: mRNA-1273 Plus Placebo
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Dose A: mRNA-1073 Plus Placebo; Dose B: mRNA-1073 Plus Placebo; Dose C: mRNA-1073 Plus Placebo; mRNA-1010 Plus Placebo; mRNA-1273 Plus Placebo

SUMMARY:
The primary goal of this study is to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1073 compared to co-administered mRNA-1010 and mRNA-1273 vaccines and to the individual vaccines alone in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18 kilograms per meter squared (kg/m^2) to 35 kg/m^2 (inclusive) at the Screening Visit.
* Participants must have been fully vaccinated for COVID-19 primary series according to the locally authorized or approved regimen, and their last COVID-19 vaccine (primary series or booster) was ≥ 120 days prior to the randomization visit (or less per local guidance).

Exclusion Criteria:

* Participant is acutely ill or febrile (temperature ≥ 38.0℃ [100.4°F]) 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day Screening window and will retain their initially assigned participant number.
* Participant has a history of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures. Clinically unstable is defined as a diagnosis or condition requiring significant changes in management or medication ≤ 60 days prior to Screening and includes ongoing workup of an undiagnosed illness that could lead to a new diagnosis or condition. Asymptomatic conditions and conditions with no evidence of end organ involvement (for example, mild hypertension, dyslipidemia) are not exclusionary, provided that they are being appropriately managed and are clinically stable (for example, unlikely to result in symptomatic illness within the time course of this study). Illnesses or conditions may be exclusionary, even if otherwise stable, due to therapies used to treat them (for example, immune-modifying treatments), at the discretion of the investigator.
* Participant has a reported history of congenital or acquired immunodeficiency, immunosuppressive condition, or immune-mediated disease.
* Participant has dermatologic conditions that could affect local solicited adverse reaction (AR) assessments (for example, tattoos, psoriasis patches affecting skin over the deltoid areas).
* Participant has a reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA vaccine(s) or any components of the mRNA vaccines.
* Participant has a reported history of bleeding disorder that is considered a contraindication to IM injection or phlebotomy.
* Participant has a diagnosis of malignancy within previous 10 years (excluding nonmelanoma skin cancer).
* Participant has any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to Screening (for corticosteroids ≥ 10 mg/day of prednisone or equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study. Inhaled, nasal, topical steroids are not exclusionary.
* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤ 28 days prior to study injections (Day 1) or plans to receive a vaccine authorized or approved by a local health agency within 28 days before or after the study injections.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine ≤ 180 days prior to the randomization visit.
* Participant has tested positive for influenza by local health authority approved testing methods ≤ 180 days prior to the Screening Visit.
* Participant has had close contact to someone with SARS-CoV-2 infection or COVID-19 as defined by the US CDC in the past 10 days prior to the Screening Visit.
* Participant has known history of SARS-CoV-2 infection within ≤ 90 days.
* Participant has received systemic immunoglobulins or blood products ≤ 90 days prior to the Screening Visit or plans to receive systemic immunoglobulins or blood products during the study.
* Participant has a history of myocarditis, pericarditis, or myopericarditis.
* Participant has donated ≥ 450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.
* Participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.
* Participant is an immediate family member or household member of study personnel, study site staff, or Sponsor personnel.

Phase 1 Specific Exclusion Criteria:

* Participant has clinical screening laboratory values (total white blood cell count, hemoglobin, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, alkaline phosphatase, and total bilirubin) > Grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Research Centers of America, Hollywood, Florida
  - AES - DRS - Optimal Research Illinois - Peoria, Peoria, Illinois
  - Meridian, Sioux City, Iowa
  - Benchmark Research, Metairie, Louisiana
  - Meridian, Norfolk, Nebraska
  - Meridian, Binghamton, New York
  - Rochester Clinical Research Inc, Rochester, New York
  - Meridian, Cincinnati, Ohio
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research - CyFair, Houston, Texas
  - DM Clinical Research - TCDD, Houston, Texas
  - J Lewis Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Rudman Spergel AK, Henry C, Nachbagauer R, Kaplonek P, Astley E, Avanesov A, Bertera H, Carmona L, Cizmeci D, Collins A, Embry A, Guo R, Mao X, Pucci A, Shao S, Shih-Lu-Lee J, Yu WH, Brune D, Chu L, Irfan M, Alter G, Ananworanich J, Shaw CA. Phase 1/2 randomized, observer-blind clinical trial of a first-generation, mRNA-based vaccine against seasonal influenza and COVID-19 in healthy adults. Hum Vaccin Immunother. 2026 Dec;22(1):2589644. doi: 10.1080/21645515.2025.2589644. Epub 2026 Feb 2. PMID 41627968
- [Derived] Sanchez-Martinez ZV, Alpuche-Lazcano SP, Stuible M, Akache B, Renner TM, Deschatelets L, Dudani R, Harrison BA, McCluskie MJ, Hrapovic S, Blouin J, Wang X, Schuller M, Cui K, Cho JY, Durocher Y. SARS-CoV-2 spike-based virus-like particles incorporate influenza H1/N1 antigens and induce dual immunity in mice. Vaccine. 2024 Dec 2;42(26):126463. doi: 10.1016/j.vaccine.2024.126463. Epub 2024 Oct 30. PMID 39481241

RESULTS

PARTICIPANT FLOW:
Groups:
- mRNA-1273 + Placebo: On Day 1, participants received 2 co-administered intramuscular (IM) injections, mRNA-1273 administered in one arm and placebo matched to mRNA-1273 in the other arm.
- mRNA-1010 + Placebo: On Day 1, participants received 2 co-administered IM injections, mRNA-1010 administered in one arm and placebo matched to mRNA-1010 in the other arm.
- mRNA-1010 + mRNA-1273: On Day 1, participants received 2 co-administered IM injections, mRNA-1010 administered in one arm and mRNA-1273 in the other arm.
- Dose A: mRNA-1073 Low Dose + Placebo: On Day 1, participants received 2 co-administered IM injections, mRNA-1073 low dose administered in one arm and placebo matched to mRNA-1073 in the other arm.
- Dose B: mRNA-1073 Medium Dose + Placebo: On Day 1, participants received 2 co-administered IM injections, mRNA-1073 medium dose administered in one arm and placebo matched to mRNA-1073 in the other arm.
- Dose C: mRNA-1073 High Dose + Placebo: On Day 1, participants received 2 co-administered IM injections, mRNA-1073 high dose administered in one arm and placebo matched to mRNA-1073 in the other arm.
Period: Overall Study
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Started | 50 | 99 | 101 | 100 | 100 | 100
Received at Least 1 Dose of Study Drug | 49 | 99 | 101 | 100 | 98 | 100
Completed | 46 | 90 | 98 | 93 | 94 | 96
Not Completed | 4 | 9 | 3 | 7 | 6 | 4
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 7 | 0 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Full analysis set consisted of all randomly assigned participants who received the investigational product (IP). Participants were analyzed according to the group to which they were randomized.
Groups:
- mRNA-1273 + Placebo: On Day 1, participants received 2 co-administered IM injections, mRNA-1273 administered in one arm and placebo matched to mRNA-1273 in the other arm.
- Total: Total of all reporting groups
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo | Total
Number analyzed (Participants) | 49 | 99 | 101 | 100 | 98 | 100 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.37) | 47.4 (14.49) | 48.5 (14.55) | 49.3 (15.10) | 49.0 (13.93) | 48.2 (14.54) | 48.4 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 54 | 65 | 55 | 56 | 64 | 323
  Male | 20 | 45 | 36 | 45 | 42 | 36 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 11 | 14 | 11 | 8 | 7 | 54
  Not Hispanic or Latino | 42 | 88 | 85 | 88 | 88 | 92 | 483
  Unknown or Not Reported | 4 | 0 | 2 | 1 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 1 | 0 | 3
  Asian | 0 | 2 | 5 | 3 | 4 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 11 | 13 | 8 | 17 | 16 | 13 | 78
  White | 37 | 83 | 85 | 79 | 76 | 83 | 443
  More than one race | 0 | 0 | 2 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reaction (ARs)
Description: Solicited ARs (local and systemic) were collected in the electronic diary (eDiary). Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. Note, that not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of all serious AEs (SAEs) and all nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to Day 8 (7 days post vaccination)
Population: The solicited safety set consisted of all participants in the safety set who contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 49 | 98 | 101 | 100 | 98 | 100
Participants
  Solicited Local ARs | 38 | 80 | 90 | 92 | 76 | 78
  Solicited Systemic ARs | 31 | 70 | 87 | 80 | 63 | 67

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent AE (TEAE) was defined as any event not present before exposure to vaccine or any event already present that worsens in intensity or frequency after exposure. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsens from baseline and is considered clinically significant in the medical and scientific judgment of the Investigator. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study, regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Day 29 (28 days post vaccination)
Population: The safety set consisted of all randomly assigned participants who received the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 49 | 99 | 101 | 100 | 98 | 100
Participants | 7 | 21 | 14 | 19 | 11 | 22

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), Medically-Attended AEs (MAAEs) and AEs Leading to Discontinuation
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner. This would include visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or COVID-19 and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to Day 181
Population: The safety set consisted of all randomly assigned participants who received the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 49 | 99 | 101 | 100 | 98 | 100
Participants
  SAEs | 2 | 1 | 0 | 0 | 1 | 0
  AESIs | 0 | 2 | 0 | 1 | 0 | 1
  MAAEs | 13 | 38 | 32 | 34 | 34 | 44
  AEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Geometric Mean Titer of Anti-Hemagglutinin Antibodies at Day 29, as Measured by Hemagglutination Inhibition Assay (HAI) For Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included BV and BY.
Time Frame: Day 29
Population: Per protocol set consisted of all participants in the FAS who comply with injection schedule, comply with timings of immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment and a Day 29 assessment, do not have influenza or SARS-CoV-2 infection at baseline and post-baseline up to Day 29 and have no major protocol deviations and/or prohibited concomitant medication use that are prespecified with impacts on immune response. N=number evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 87 | 94 | 91 | 86 | 95
titer
  Influenza A H1N1 Antibody | 175.41 [139.67 to 220.30] | 134.04 [110.72 to 162.26] | 104.78 [82.94 to 132.39] | 111.33 [90.94 to 136.29] | 108.68 [88.64 to 133.26]
  Influenza A H3N2 Antibody | 189.9 [145.67 to 247.54] | 214.12 [171.36 to 267.56] | 144.36 [111.87 to 186.29] | 141.15 [112.68 to 176.80] | 129.94 [103.77 to 162.715]
  Influenza B BV Antibody | 106.22 [89.66 to 125.83] | 107.91 [92.79 to 125.50] | 91.78 [77.16 to 109.16] | 89.27 [75.92 to 104.98] | 84.82 [72.56 to 99.15]
  Influenza B BY Antibody | 194.51 [163.21 to 231.81] | 182.01 [152.26 to 217.58] | 139.48 [112.70 to 172.61] | 130.27 [107.67 to 157.61] | 121.29 [99.73 to 147.52]

5. Secondary Outcome: Geometric Mean Titer of VAC62 Neutralizing Antibody at Day 29, as Measured by Pseudovirus Neutralization Assay (or Binding Antibody Assay) For Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 43 | 93 | 88 | 85 | 92
titer | 8477.30 [6424.05 to 11186.62] | 6075.76 [5119.62 to 7210.47] | 7573.97 [6475.43 to 8858.86] | 5678.54 [4671.74 to 6902.32] | 4410.29 [3762.65 to 5169.41]

6. Secondary Outcome: Geometric Mean Fold Rise of Anti-Hemagglutinin Antibodies at Day 29, as Measured by Hemagglutination Inhibition Assay (HAI) For Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included BV and BY.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 87 | 94 | 91 | 86 | 95
ratio
  Influenza A H1N1 Antibody | 3.97 [3.19 to 4.95] | 3.31 [2.76 to 3.96] | 2.25 [1.89 to 2.68] | 2.48 [2.06 to 2.98] | 2.67 [2.21 to 3.23]
  Influenza A H3N2 Antibody | 5.82 [4.56 to 7.43] | 5.07 [4.19 to 6.14] | 3.84 [3.22 to 4.58] | 4.15 [3.33 to 5.18] | 3.41 [2.80 to 4.14]
  Influenza B BV Antibody | 1.61 [1.42 to 1.82] | 1.64 [1.47 to 1.84] | 1.29 [1.14 to 1.44] | 1.29 [1.18 to 1.43] | 1.29 [1.16 to 1.43]
  Influenza B BY Antibody | 2.68 [2.25 to 3.19] | 2.17 [1.85 to 2.53] | 1.63 [1.46 to 1.83] | 1.65 [1.46 to 1.87] | 1.58 [1.41 to 1.78]

7. Secondary Outcome: Geometric Mean Fold Rise of VAC62 Neutralizing Antibody at Day 29, as Measured by Pseudovirus Neutralization Assay (or Binding Antibody Assay) For SARS-CoV-2
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. 95% CI was calculated based on the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 43 | 93 | 88 | 85 | 92
ratio | 6.14 [3.98 to 9.48] | 4.07 [3.26 to 5.07] | 3.50 [2.76 to 4.44] | 3.45 [2.82 to 4.22] | 3.18 [2.73 to 3.69]

8. Secondary Outcome: Percentage of Participants With Seroconversion as Measured by HAI Assay For Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seroconversion at a participant level is defined as a pre-vaccination HAI titer < 1:10 and a post-vaccination HAI titer >= 1:40 or a pre-vaccination HAI titer >= 1:10 and a minimum 4-fold rise in post vaccination HAI antibody titer.
Time Frame: Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 87 | 94 | 91 | 86 | 95
percentage of participants
  Influenza A H1N1 Antibody | 47.1 [36.3 to 58.1] | 42.6 [32.4 to 53.2] | 27.5 [18.6 to 37.8] | 31.4 [21.8 to 42.3] | 31.6 [22.4 to 41.9]
  Influenza A H3N2 Antibody | 64.4 [53.4 to 74.4] | 63.8 [53.3 to 73.5] | 53.8 [43.1 to 64.4] | 53.5 [42.4 to 64.3] | 42.1 [32.0 to 52.7]
  Influenza B BV Antibody | 16.1 [9.1 to 25.5] | 9.6 [4.5 to 17.4] | 3.3 [0.7 to 9.3] | 2.3 [0.3 to 8.1] | 6.3 [2.4 to 13.2]
  Influenza B BY Antibody | 32.2 [22.6 to 43.1] | 19.1 [11.8 to 28.6] | 11.0 [5.4 to 19.3] | 10.5 [4.9 to 18.9] | 10.5 [5.2 to 18.5]

9. Secondary Outcome: Percentage of Participants With Seroresponse as Measured by PsVNA (or Binding Antibody Assay) For SARS-CoV-2
Description: Seroresponse at a participant level is defined as an increase from below the lower limit of quantification (LLOQ) to >= 4 x LLOQ if baseline neutralizing antibody (nAb) level is < LLOQ, or >= 4 fold rise if baseline nAb level is >=LLOQ.
Time Frame: Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
Number analyzed (Participants) | 43 | 93 | 88 | 85 | 92
percentage of participants | 52.4 [36.4 to 68.0] | 44.4 [34.0 to 55.3] | 37.5 [27.4 to 48.5] | 36.5 [26.3 to 47.6] | 35.9 [26.1 to 46.5]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 181
Description: The safety set consisted of all randomly assigned participants who received the IP. Participants will be included in the vaccination group corresponding to what they actually received. Note, that not all solicited ARs were considered AEs. The Investigator reviewed whether the solicited AR was also to be recorded as an AE.
Arm/Group | mRNA-1273 + Placebo | mRNA-1010 + Placebo | mRNA-1010 + mRNA-1273 | Dose A: mRNA-1073 Low Dose + Placebo | Dose B: mRNA-1073 Medium Dose + Placebo | Dose C: mRNA-1073 High Dose + Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/99 | 0/101 | 0/100 | 0/98 | 0/100
Serious Adverse Events (participants affected / at risk) | 2/49 | 1/99 | 0/101 | 0/100 | 1/98 | 0/100
Other Adverse Events (participants affected / at risk) | 42/49 | 86/99 | 93/101 | 94/100 | 81/98 | 89/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mRNA-1273 + Placebo (N=49) | mRNA-1010 + Placebo (N=99) | mRNA-1010 + mRNA-1273 (N=101) | Dose A: mRNA-1073 Low Dose + Placebo (N=100) | Dose B: mRNA-1073 Medium Dose + Placebo (N=98) | Dose C: mRNA-1073 High Dose + Placebo (N=100)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mRNA-1273 + Placebo (N=49) | mRNA-1010 + Placebo (N=99) | mRNA-1010 + mRNA-1273 (N=101) | Dose A: mRNA-1073 Low Dose + Placebo (N=100) | Dose B: mRNA-1073 Medium Dose + Placebo (N=98) | Dose C: mRNA-1073 High Dose + Placebo (N=100)
COVID-19 (Infections and infestations) | 3 | 14 | 11 | 13 | 13 | 18
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 1 | 3 | 8 | 11
Rhinovirus infection (Infections and infestations) | 1 | 4 | 9 | 2 | 8 | 4
Headache (Nervous system disorders) | 18 | 41 | 64 | 63 | 42 | 45
Vomiting (Gastrointestinal disorders) | 7 | 14 | 23 | 14 | 14 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 52 | 73 | 59 | 42 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 30 | 49 | 49 | 35 | 31
Injection site pain (General disorders) | 38 | 80 | 89 | 91 | 76 | 78
Fatigue (General disorders) | 25 | 57 | 79 | 67 | 45 | 51
Chills (General disorders) | 10 | 31 | 51 | 46 | 30 | 20
Injection site lymphadenopathy (General disorders) | 15 | 19 | 25 | 26 | 20 | 22
Pyrexia (General disorders) | 2 | 4 | 20 | 17 | 5 | 2
Injection site induration (General disorders) | 6 | 2 | 4 | 10 | 3 | 4
Injection site erythema (General disorders) | 0 | 0 | 2 | 8 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT05375838/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT05375838/SAP_001.pdf